CLINICAL TRIAL: NCT05338593
Title: Therapy and Outcome of Prolonged Veno-venous ECMO Therapy of Critically Ill ARDS Patients.
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Armin N. Flinspach, Principal Investigator, Goethe University
Other Study IDs: prolonged VV-ECMO
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; Outcome, Fatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- prolonged veno-venous extracorporeal membrane oxygenation: Critically affected patients treated with veno-venous extracorporeal membrane oxygenation (VV-ECMO). Based on severe acute respiratory distress syndrome (ARDS) and prolonged therapy for more than 2 weeks.
  Interventions: Other: Outcome

INTERVENTIONS:
Other: Outcome — Mortality rate of prolonged therapy.

SUMMARY:
In the context of the coronavirus (COVID-19) pandemic, healthcare systems worldwide faced an unprecedented shortage of severe ARDS. Critically affected patients were treated with veno-venous extracorporeal membrane oxygenation (VV-ECMO) for complete respiratory failure early in the pandemic. Due to a shortage of resources in the sense of terminal equipment and adequately trained personnel with appropriate expertise in many countries and regions, a strict selection of suitable patients was made. Repeatedly, it was observed that patients under VV-ECMO also needed several weeks to recover sufficiently to generate device sufficient gas exchange. Due to the scarcity of VV-ECMO resources outside of the pandemic, the question arose whether a prolonged therapy still holds a sufficient prospect of success and what the course of treatment of such patients would be like.

ELIGIBILITY:
Inclusion Criteria:

veno-venous extracorporeal membrane oxygenation

Exclusion Criteria:

veno-arterial extracorporeal membrane oxygenation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically affected patients treated with veno-venous extracorporeal membrane oxygenation (VV-ECMO). Based on severe acute respiratory distress syndrome (ARDS) and prolonged therapy for more than 2 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Mortality | During intensive care treatment (Usually within 25 weeks)
  Mortality rate under ongoing veno-venous extracorporeal membrane oxygenation over time

SECONDARY OUTCOMES:
Major bleeding | During intensive care treatment (Usually within 25 weeks)
  Number of patients with critical bleeding events during therapy, needing red blood cell transfusion
critical device error | During intensive care treatment (Usually within 25 weeks)
  Number of patients with a critical device errors of the veno-venous extracorporeal membrane oxygenation device.

CONTACTS AND LOCATIONS:
Overall Officials: Armin N Flinspach, M.D., Principal Investigator — JWGoethe University
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No
Sharing patient data is not possible due to national and local legal restrictions.